CLINICAL TRIAL: NCT04818411
Title: Comparison of Stabilization Exercises Versus Thrust Manipulation Technique on Pelvic Girdle Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-UOL-FAHS/659 Anam Naz
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Pelvic Girdle Pain
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine physical therapy treatment with the Stabilization exercises (Active Comparator): Stabilization exercises
  Interventions: Other: Routine physical therapy treatment with the Stabilization exercises
- Routine physical therapy treatment + High-velocity thrust manipulation (Experimental): High-velocity thrust manipulation
  Interventions: Other: Routine physical therapy treatment + High-velocity thrust manipulation

INTERVENTIONS:
Other: Routine physical therapy treatment with the Stabilization exercises — The program was based on specific training of the transversely oriented abdominal muscles with coactivation of the lumbar multifidus at the lumbosacral region, training of the gluteus maximus, the latissimus dorsi, the oblique abdominal muscles, the erector spinae, the quadratus lumborum, and the hip adductors and abductors. Initially, we focused on the specific contraction of the transversely oriented abdominal muscles. After approximately 2 weeks, loading was progressively increased throughout the intervention period. The women were required to exercise for 30 to 60 minutes, 3 days a week, for 3-4 weeks.
  Arms: Routine physical therapy treatment with the Stabilization exercises
Other: Routine physical therapy treatment + High-velocity thrust manipulation — : For high-velocity thrust technique, a modified Chicago technique was used. For this procedure, the lumbopelvic region was targeted. The side to be treated was chosen, based on the subject's report of her most symptomatic side. The physical therapist, performed passively side bend the subject toward the painful side, rotate the upper body in the direction opposite to the side bending, and then deliver a quick posterior and inferior thrust at a grade V including a small-amplitude/high-velocity therapeutic movement. A maximum of 2 attempts per side was permitted if no pop was heard following the first attempt. If the subject showed improvement of 50% or less after the first treatment, the intervention was categorized as a failure, the examination and intervention were repeated, and the subjects were asked to return 2 to 4 days later. If the subject showed greater than 50% improvement, the intervention was categorized as a success, and study participation was concluded.
  Arms: Routine physical therapy treatment + High-velocity thrust manipulation

SUMMARY:
The objective of this research is to compare the efficacy of stabilization exercise versus pelvic girdle pain thrust manipulation technique in females with postpartum pain.

DETAILED DESCRIPTION:
Pelvic-girdle pain is a mechanical disorder growing rapidly as a consequence of changing delivery pattern and changing lifestyle. Medication with synthetic drugs not only has been unable to effectively curtail the spread of this disease conditions but also is most of the times linked with co-occurring side-effects. The exercise and manual therapy-based approach could lead in reducing the functional limitations and morbidity rate in females with the postpartum pain. This research could also help in spreading the awareness globally, to Prenatal and Postnatal Hospital Caregivers.

ELIGIBILITY:
Inclusion Criteria:

* • Post-partum females with the normal vaginal delivery present with pelvic girdle pain before the next conception.

  * Aged between 18 and 45
  * Posterior pelvic girdle pain located distal and/or lateral to the L5-S1
  * Pain onset during pregnancy or within 3 weeks after delivery, most recent delivery within 6 to 16 weeks
  * Positive posterior pelvic pain provocation (P4) test

Exclusion Criteria:

* Patients presenting with the history of:

  * Back pain indicating radiculopathy
  * Mechanical back pain
  * Back pain due to disc herniation
  * Rheumatological diseases
  * Neurological illness or recent surgery
  * Women who have gone through C-section

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-08-18 (Actual); Primary Completion 2020-06-27 (Actual); Study Completion 2020-07-26 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 2 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Oswestry disability index | 2 months
  The ODI score (index) is calculated as: If all 10 sections are completed the score is calculated as follows: if 16 (total scored) out of 50 (total possible score) x 100 = 32% If one section is missed (or not applicable) the score is calculated: If 16 (total scored) / 45 (total possible score) x 100 = 35.5%

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bastiaanssen JM, de Bie RA, Bastiaenen CH, Essed GG, van den Brandt PA. A historical perspective on pregnancy-related low back and/or pelvic girdle pain. Eur J Obstet Gynecol Reprod Biol. 2005 May 1;120(1):3-14. doi: 10.1016/j.ejogrb.2004.11.021. PMID 15866079
- [Background] Bergstrom C, Persson M, Mogren I. Sick leave and healthcare utilisation in women reporting pregnancy related low back pain and/or pelvic girdle pain at 14 months postpartum. Chiropr Man Therap. 2016 Feb 15;24:7. doi: 10.1186/s12998-016-0088-9. eCollection 2016. PMID 26885363
- [Background] Vermani E, Mittal R, Weeks A. Pelvic girdle pain and low back pain in pregnancy: a review. Pain Pract. 2010 Jan-Feb;10(1):60-71. doi: 10.1111/j.1533-2500.2009.00327.x. Epub 2010 Oct 26. PMID 19863747
- [Background] Robinson HS, Eskild A, Heiberg E, Eberhard-Gran M. Pelvic girdle pain in pregnancy: the impact on function. Acta Obstet Gynecol Scand. 2006;85(2):160-4. doi: 10.1080/00016340500410024. PMID 16532908
- [Background] Bergstrom C, Persson M, Nergard KA, Mogren I. Prevalence and predictors of persistent pelvic girdle pain 12 years postpartum. BMC Musculoskelet Disord. 2017 Sep 16;18(1):399. doi: 10.1186/s12891-017-1760-5. PMID 28915804
- [Background] Eggen MH, Stuge B, Mowinckel P, Jensen KS, Hagen KB. Can supervised group exercises including ergonomic advice reduce the prevalence and severity of low back pain and pelvic girdle pain in pregnancy? A randomized controlled trial. Phys Ther. 2012 Jun;92(6):781-90. doi: 10.2522/ptj.20110119. Epub 2012 Jan 26. PMID 22282770